CLINICAL TRIAL: NCT06657443
Title: The Effect of a Peer Mentoring Program on Nursing Students' Perceived Empathic Self-Efficacy, Social Self-Efficacy, and Youth Leadership Characteristics: A Pretest-Posttest Quasi-Experimental Study
Brief Title: The Effect of a Peer Mentoring Program on Nursing Students
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, TANGÜL AYTUR ÖZEN, Dr, Asst. Prof. Dr., Head of the Department of Nursing Management, Principal Investigator., Suleyman Demirel University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: SDU-SBF-HEM-TAO-01
Record Dates: First submitted 2024-10-22; First posted 2024-10-24 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Peer Group; Mentoring; Program Evaluation; Nurse; Empathy Skills; Social Skills; Leadership
Keywords: Peer mentoring program; Nursing students,; Empathic Self-Efficacy; Social Self-Efficacy; Youth Leadership
MeSH Terms: conditions — Social Skills

STUDY DESIGN:
Masking Description: The two researchers involved in the study will contact the mentee students who have enrolled at the beginning of the autumn term of the 2024-2025 academic year and make the assignments of the peer mentors. These processes will be carried out by an independent researcher. Peer mentor and mentee assignments will remain confidential from the researchers until the pre-test is conducted by the research team.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Training material sharing and activity sessions (Experimental): Eğitim materyali paylaşımı ve etkinlik oturumları
  Interventions: Other: First Session; Other: Second Session; Other: Third session; Other: Fourth session; Other: Fifth Session; Other: Sixth Session

INTERVENTIONS:
Other: First Session — Introductions, explanation of the purpose and content of the project, realisation of the pre-test application. Giving the assignment with the theme of 'Nursing and Society' between peer mentors and mentees.
Other: Second Session — Training of peer mentors on communication techniques, interview methods and empathic approach.
Other: Third session — Sharing postcasts on communication techniques, interview methods and empathic approach with peer mentors.
Other: Fourth session — Training of peer mentors on social motivation and leader-member interaction
Other: Fifth Session — Sharing postcasts with peer mentors on social motivation and leader-member interaction.
Other: Sixth Session — Presentation of 'Nursing and Society' themed assignments of peer mentors and mentees as a group (Composition, poem, poster, presentation, role play, etc. are left free among the students) and post-test application.

SUMMARY:
This project is designed as a quasi-experimental study to evaluate the effect of the Peer Leadership Program, established in the Nursing Department, on nursing peer mentor students' empathic self-efficacy, social self-efficacy, and youth leadership characteristics.

DETAILED DESCRIPTION:
The study population comprises second, third and fourth-year students enrolled at Süleyman Demirel University, Faculty of Health Sciences, Department of Nursing, during the 2024-2025 academic year. Peer mentor students, selected on the basis of volunteerism, will be randomly assigned mentors by an independent researcher to ensure randomness. The study will be conducted over a period of six weeks. During this period, the peer mentors will undergo training in communication techniques, interview methods, empathic approach, social motivation and leader-member interaction, with the subsequent sharing of postcasts. Furthermore, a presentation and evaluation meeting will be held between the peer mentors and their mentees, with the aim of fostering empathy and understanding between the two groups. The meeting will be based on the theme of 'nursing and society'. In order to assess the effectiveness of the intervention, the peer mentors' empathic self-efficacy, social self-efficacy and youth leadership characteristics will be evaluated before and after the meeting. Additionally, the socio-demographic data of the students will be recorded in a data collection form.

ELIGIBILITY:
Inclusion Criteria:

* The term "volunteers" is used to designate students enrolled in the 2024-2025 academic year, in their second, third or fourth year of studies, who are actively engaged in the education and training process.

Exclusion Criteria:

* Students who indicated a preference for not being a first-year student and instead volunteered to serve as peer mentors.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-10-29 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-04-24 (Estimated)

PRIMARY OUTCOMES:
Perceived Empathic Self-Efficacy and Social Self-Efficacy Scale | Before Training and Activities (First Session) and at the Final Session After 6 Weeks
  The scale was developed by Di Giunta et al. (2010), and the Turkish validity and reliability study was conducted by Akın and Başören. The scale comprises 11 items and two dimensions, with respondents invited to indicate their level of agreement on a five-point Likert scale, where 1 represents a complete disagreement and 5 represents complete agreement. The items are distributed according to the two subscales, namely perceived empathic self-efficacy (items 1-6) and perceived social self-efficacy (items 7-11). A high score on the first sub-dimension of the scale, empathic self-efficacy, indicates that the individual perceives themselves as capable of responding empathically to the needs and feelings of others. A high score on the second sub-dimension, social self-efficacy, indicates that the individual perceives themselves as capable of initiating and managing interpersonal relationships.

SECONDARY OUTCOMES:
Youth Leadership Traits scale | Before Training and Activities (First Session) and at the Final Session After 6 Weeks
  The 'Youth Leadership Characteristics Scale' developed by Cansoy and Turan in 2016 in 5-point Likert form consists of 40 items and seven sub-dimensions.
  The sub-dimensions are; willingness to struggle and goal setting (7 items), ability to communicate (7 items), group skills (7 items), decision making skills (4 items), problem solving skills (4 items), responsibility (5 items), self-confidence (6 items). In Cansoy and Turan's (2016) study, the Cronbach's Alpha value of the scale was found to be 0.92. According to the frequency of the behaviour shown, the youth leadership traits scale is planned as Always '5 points', Frequently '4 points', Occasionally '3 points', Very rarely '2 points', Never '1 point'. The increase in the score indicates that the approach is positive.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Suleyman Demirel University — https://w3.sdu.edu.tr/